CLINICAL TRIAL: NCT01576575
Title: Influence of CYP3A Modulation on Buprenorphine Disposition and Clinical Effects
Brief Title: Buprenorphine Disposition and CYP3A
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: 201104146
Record Dates: First submitted 2012-04-10; First posted 2012-04-12 (Estimated); Results first posted 2020-01-22 (Actual); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: Healthy
Keywords: buprenorphine CYP3A
MeSH Terms: interventions — Buprenorphine; Rifampin; Ketoconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Healthy males and non-pregnant females (Experimental): Subjects will be studied during a maximum of seven occasions.
  Study drugs are intravenous buprenorphine (0.025-0.2 mg infused over 1 hr) and sublingual buprenorphine (2-4 mg), with 1-3 week washout between sessions.
  Sessions 1&2: Control (no pretreatment) - intravenous and sublingual buprenorphine. Some subjects will only undergo session 1 (IV)
  Sessions 3&4: Liver and gut CYP3A induction (rifampin 600 mg daily), intravenous and sublingual buprenorphine
  Session 5: Gut only CYP3A inhibition (grapefruit juice the night before), sublingual buprenorphine
  Sessions 6&7: Liver and gut CYP3A inhibition (ketoconazole 400 mg daily), intravenous and sublingual buprenorphine
  Interventions: Drug: Buprenorphine Control; Drug: Buprenorphine + Rifampin; Drug: Buprenorphine + Grapefruit juice; Drug: Buprenorphine + Ketoconazole

INTERVENTIONS:
Drug: Buprenorphine Control — Control (no pretreatment) - intravenous and sublingual buprenorphine. Some subjects will only undergo session 1 (IV)
Drug: Buprenorphine + Rifampin — Liver and gut CYP3A induction (rifampin 600 mg daily), intravenous and sublingual buprenorphine
Drug: Buprenorphine + Grapefruit juice — Gut only CYP3A inhibition (grapefruit juice the night before), sublingual buprenorphine
Drug: Buprenorphine + Ketoconazole — Liver and gut CYP3A inhibition (ketoconazole 400 mg daily), intravenous and sublingual buprenorphine

SUMMARY:
To evaluate role of CYP3A in buprenorphine disposition and effect

DETAILED DESCRIPTION:
Subjects will be studied during a maximum of seven occasions.

Study drugs are intravenous buprenorphine (0.025-0.2 mg infused over 1 hr) and sublingual buprenorphine (2-4 mg), with 1-3 week washout between sessions.

Sessions 1&2: Control (no pretreatment) - intravenous and sublingual buprenorphine. Some subjects will only undergo session 1 (IV)

Sessions 3&4: Liver and gut CYP3A induction (rifampin 600 mg daily), intravenous and sublingual buprenorphine

Session 5: Gut only CYP3A inhibition (grapefruit juice the night before), sublingual buprenorphine

Sessions 6&7: Liver and gut CYP3A inhibition (ketoconazole 400 mg daily), intravenous and sublingual buprenorphine

ELIGIBILITY:
Inclusion Criteria:

Each subject must meet all of the following criteria:

1. Male or non-pregnant female volunteer, 18-50 yr old
2. Good general health with no known major medical conditions
3. BMI < 33
4. Provide informed consent

Exclusion Criteria:

Subjects will not be enrolled if any of the following criteria exist:

1. Known history of liver or kidney disease
2. Use of prescription or non-prescription medications, herbals or foods known to be metabolized by or affect CYP3A activity (this includes the use of oral contraceptives).
3. Females who are pregnant or nursing
4. Known history of drug or alcohol addiction (prior or present addiction or addiction treatment)
5. Direct physical access to and routine handling of addicting drugs in the regular course of duty (this is a routine exclusion from studies of drugs with addiction potential)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2010-06; Primary Completion 2014-03-29 (Actual); Study Completion 2014-03-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Evan Kharasch, MD, PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- [Background] Heel RC, Brogden RN, Speight TM, Avery GS. Buprenorphine: a review of its pharmacological properties and therapeutic efficacy. Drugs. 1979 Feb;17(2):81-110. doi: 10.2165/00003495-197917020-00001. PMID 378645
- [Background] Pickworth WB, Johnson RE, Holicky BA, Cone EJ. Subjective and physiologic effects of intravenous buprenorphine in humans. Clin Pharmacol Ther. 1993 May;53(5):570-6. doi: 10.1038/clpt.1993.72. PMID 8491067
- [Background] Walsh SL, Preston KL, Bigelow GE, Stitzer ML. Acute administration of buprenorphine in humans: partial agonist and blockade effects. J Pharmacol Exp Ther. 1995 Jul;274(1):361-72. PMID 7542336

RESULTS

PARTICIPANT FLOW:
Groups:
- Healthy Volunteers: Healthy males and non-pregnant females
Period: Buprenorphine Control
Arm/Group | Healthy Volunteers
Started | 21
Completed | 18
Not Completed | 3
Not completed — Withdrawal by Subject | 3
Period: Buprenorphine + Rifampin
Arm/Group | Healthy Volunteers
Started | 18
Completed | 15
Not Completed | 3
Not completed — Withdrawal by Subject | 3
Period: Buprenorphine + Grapefruit
Arm/Group | Healthy Volunteers
Started | 15
Completed | 14
Not Completed | 1
Not completed — Withdrawal by Subject | 1
Period: Buprenorphine + Ketoconazole
Arm/Group | Healthy Volunteers
Started | 14
Completed | 14
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Healthy Volunteers: Subjects will be studied during a maximum of seven occasions.
  Study drugs are intravenous buprenorphine (0.025-0.2 mg infused over 1 hr) and sublingual buprenorphine (2-4 mg), with 1-3 week washout between sessions.
  Sessions 1&2: Control (no pretreatment) - intravenous and sublingual buprenorphine. Some subjects will only undergo session 1 (IV)
  Sessions 3&4: Liver and gut CYP3A induction (rifampin 600 mg daily), intravenous and sublingual buprenorphine
  Session 5: Gut only CYP3A inhibition (grapefruit juice the night before), sublingual buprenorphine
  Sessions 6&7: Liver and gut CYP3A inhibition (ketoconazole 400 mg daily), intravenous and sublingual buprenorphine
Arm/Group | Healthy Volunteers
Number analyzed (Participants) | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 27 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 13

OUTCOME MEASURES:

1. Primary Outcome: Plasma Cmax of Buprenorphine
Time Frame: 96 hr
Population: 0 participants analyzed. The PI has left the institution. Sincere efforts were made to contact the PI but were unsuccessful. No study data are available.
Groups:
- Control (no Pretreatment): Sessions 1&2: Control (no pretreatment) - intravenous and sublingual buprenorphine. Some subjects will only undergo session 1 (IV)
- Rifampin: Sessions 3&4: Liver and gut CYP3A induction (rifampin 600 mg daily), intravenous and sublingual buprenorphine
- Grapefruit Juice: Session 5: Gut only CYP3A inhibition (grapefruit juice the night before), sublingual buprenorphine
- Ketoconazole: Sessions 6&7: Liver and gut CYP3A inhibition (ketoconazole 400 mg daily), intravenous and sublingual buprenorphine
Arm/Group | Control (no Pretreatment) | Rifampin | Grapefruit Juice | Ketoconazole
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 96 hours following dosing
Groups:
- Liver and Gut CYP3A Induction: Sessions 3&4: Liver and gut CYP3A induction (rifampin 600 mg daily), intravenous and sublingual buprenorphine
- Gut Only CYP3A Inhibition: Session 5: Gut only CYP3A inhibition (grapefruit juice the night before), sublingual buprenorphine
- Liver and Gut CYP3A Inhibition: Sessions 6&7: Liver and gut CYP3A inhibition (ketoconazole 400 mg daily), intravenous and sublingual buprenorphine
Arm/Group | Control (no Pretreatment) | Liver and Gut CYP3A Induction | Gut Only CYP3A Inhibition | Liver and Gut CYP3A Inhibition
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/18 | 0/14 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/18 | 0/14 | 0/13
Other Adverse Events (participants affected / at risk) | 21/21 | 15/18 | 14/14 | 13/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control (no Pretreatment) (N=21) | Liver and Gut CYP3A Induction (N=18) | Gut Only CYP3A Inhibition (N=14) | Liver and Gut CYP3A Inhibition (N=13)
nausea (Gastrointestinal disorders) | 12 (40) | 13 (39) | 11 (21) | 12 (30) — Adverse Event Reporting Description by Arms/Groups are combined as individual results not available. Adverse events all due to buprenorphine not pretreatments
itch (General disorders) | 14 (32) | 10 (32) | 11 (16) | 8 (25) — Adverse Event Reporting Description by Arms/Groups are combined as individual results not available. Adverse events all due to buprenorphine not pretreatments
Headache (Nervous system disorders) | 4 (6) | 2 (3) | 3 (5) | 5 (15)
Dizzyness (Nervous system disorders) | 4 (15) | 3 (7) | 1 (2) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes